CLINICAL TRIAL: NCT04211493
Title: Empowering Health: Acute Psychological Effects of a Single Electromyostimulation-Whole-Body-Workout in Participants With Depression
Brief Title: Empowering Health: Acute Psychological Effects of an Electromyostimulation-Whole-Body-Workout
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Sonnenfeld-Stiftung (Unknown); Robert-Enke-Stiftung (Unknown); miha bodytec GmbH (Unknown)
Responsible Party: Principal Investigator, Antonia Bendau, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EA4/058/19
Record Dates: First submitted 2019-12-19; First posted 2019-12-26 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Depression
Keywords: Physical Activity; Physical Exercise; Mental Disorder; Depression; Mental Health; Health Behaviour; Electromyostimulation; EMS; Strength Training
MeSH Terms: conditions — Depression; Motor Activity; Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study has a randomised placebo-controlled crossover design. Every participant exercises two training-sessions (experimental-condition, placebo-condition) in randomized order with one week fade-out phase inbetween.
Who Masked: Participant
Masking Description: Participants are not aware of the study hypothesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental-Condition (Experimental): 20 minutes whole-body-workout with simultaneous muscle stimulation (EMS).
  Participants carry out easy whole-body-exercises while wearing a EMS-vest-belt-system with interwoven electrodes. During the workout the muscles are simultaneously stimulated by those external electrodes with medium level (5) of stimulation intensity.
  Interventions: Behavioral: whole-body-workout; Device: EMS
- Placebo-Condition (Placebo Comparator): 20 minutes whole-body-workout without simultaneous muscle stimulation (EMS).
  Participants carry out easy whole-body-exercises while wearing a EMS-vest-belt-system with interwoven electrodes. During the workout they are stimulated with the lowest possible stimulation intensity (1). This is perceptible as a slight tingling sensation but the impulse intensity lies below the muscular threshold and therefore generates no muscular activity.
  Interventions: Behavioral: whole-body-workout; Device: EMS-Placebo

INTERVENTIONS:
Behavioral: whole-body-workout — 20 minutes whole-body-workout
Device: EMS — Electromyostimulation-intensity 5 (muscle stimulation)
  Arms: Experimental-Condition
Device: EMS-Placebo — Electromyostimulation-intensity 1 (no muscle stimulation)
  Arms: Placebo-Condition

SUMMARY:
The study investigates the acute psychological effects of a whole-body-workout using Electromyostimulation (EMS) in participants with depression and healthy individuals.

DETAILED DESCRIPTION:
EMS-whole-body-workouts are less time-consuming and effort-intensive but generate physical effects which are comparable to conventional strength training. Therefore EMS could lower the barrier to physical activity. The present study focusses on acute psychological effects of an EMS workout - especially with regard to the reduction of depressive symptoms. Physical activity is notably important for patients with depression and shows multiple positive psychological and physical effects. But due to disease-related factors like lethargy, physical activity is far too rarely implemented. Therefore EMS-whole-body-workouts could provide an opportunity to generate positive psychological effects through a less (subjective) cost-intense strength training.

ELIGIBILITY:
Inclusion Criteria:

* Subject familiarized with experimental procedure and had given written informed consent
* Depression, according to ICD-10
* BDI-II Score ≥ 14
* Able to understand German
* Reachability of participant for the two training sessions

Exclusion Criteria:

* Contraindications for physical exercise
* Contraindications for EMS-use
* Current EMS-use
* Pregnancy
* Borderline personality disorder
* Bipolar Disorder
* Schizophrenia
* Anorexia Nervosa, Bulimia Nervosa
* Dementia
* Acute suicidality
* Substance dependencies with actual consumption (except nicotine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms | From directly before the intervention to immediately after the intervention - both: before/after the EMS-training-session and before/after the Placebo-session
  Depressive symptoms are measured using the State-Scale of the State-Trait Depression Scales (STDS) by Spaderna, Schmukle & Krohne (2002). The SDTS State-Scale has two subscales with each 5 likert scaled items with values ranging from 1 to 4. Higher scores mean a worse outcome for the first subscale and a better outcome for the second subscale.

SECONDARY OUTCOMES:
Change in anxiety symptoms | From directly before the intervention to immediately after the intervention - both: before/after the EMS-training-session and before/after the Placebo-session
  Anxiety symptoms are measured using the the State-Scale of the State-Trait Anxiety Inventory (STAI) by Laux, Glanzmann, Schaffner & Spielberger (1981). The STAI State-Scale has 20 likert scaled items with values ranging from 1 to 4, higher scores mean a worse outcome.
Change in general self-efficacy | From directly before the intervention to immediately after the intervention - both: before/after the EMS-training-session and before/after the Placebo-session
  General self-efficacy is measured using the General-Self-Efficacy Scale (GSE) by Jerusalem & Schwarzer (1981). The GSE has 10 likert scaled items with values ranging from 1 to 4, higher scores mean a better outcome.
Change in intention for physical activity | From directly before the intervention to immediately after the intervention - both: before/after the EMS-training-session and before/after the Placebo-session
  Intention for physical activity is measured using two likert scaled items by Petzold et al. (2017). Values ranging from 1 to 4, higher scores mean a better outcome.
Change in self-efficacy regarding physical activity | From directly before the intervention to immediately after the intervention - both: before/after the EMS-training-session and before/after the Placebo-session
  Self-efficacy is measured using two likert scaled items by Petzold et al. (2017). Values ranging from 1 to 4, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Ströhle, Prof.Dr., Study Director — Charité-Universitätsmedizin Berlin - Department of Psychiatry and Psychotherapy; Antonia Bendau, M.Sc.Psych., Principal Investigator — Charité-Universitätsmedizin Berlin - Department of Psychiatry and Psychotherapy
Locations (1):
- Charité-Universitätsmedizin Berlin - Department of Psychiatry and Psychotherapy, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No